CLINICAL TRIAL: NCT00445861
Title: Cetuximab in Combination With Radiation Therapy and Chemotherapy Prior to Surgery in Patients With Resectable, Locally Advanced Esophageal Carcinoma. A Multicenter Phase IB-II Trial
Brief Title: Cetuximab, Docetaxel, Cisplatin, and Radiation Therapy in Treating Patients With Locally Advanced Esophageal Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 75/06; EU-20702
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cetuximab + docetaxel + cisplatin — Chemoimmunotherapy: Patients receive cetuximab IV over 1-2 hours once weekly in weeks 1-3 and docetaxel IV over 1 hour and cisplatin IV over 1 hour once in week 1. Treatment repeats every 3 weeks for 2 courses.
Biological: Treatment level 1 — Treatment level 1: Patients receive cetuximab IV over 1 hour once weekly, cisplatin IV over 1 hour once weekly, and undergo radiotherapy once daily, 5 days a week, in weeks 7-11.
Biological: Treatment level 2 — Patients receive cetuximab, cisplatin, and radiotherapy as in treatment level 1. Patients also receive docetaxel IV over 1-2 hours once weekly in weeks 7-11.
Procedure: conventional surgery — Between 4-8 weeks after completion of neoadjuvant chemoimmunotherapy and radiotherapy, patients undergo surgery.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving cetuximab, docetaxel, and cisplatin together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I/II trial is studying the side effects of cetuximab, docetaxel, cisplatin, and radiation therapy and to see how well they work in treating patients with locally advanced esophageal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of neoadjuvant radiotherapy in combination with cetuximab, docetaxel, and cisplatin in patients with resectable locally advanced esophageal cancer.

Secondary

* Determine the feasibility and efficacy of this regimen in these patients.
* Determine the duration of response and patterns of failure in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Chemoimmunotherapy: Patients receive cetuximab IV over 1-2 hours once weekly in weeks 1-3 and docetaxel IV over 1 hour and cisplatin IV over 1 hour once in week 1. Treatment repeats every 3 weeks for 2 courses.
* Chemoimmunotherapy and radiotherapy: Patients are sequentially assigned to 1 of 2 treatment levels.

  * Treatment level 1: Patients receive cetuximab IV over 1 hour once weekly, cisplatin IV over 1 hour once weekly, and undergo radiotherapy once daily, 5 days a week, in weeks 7-11.
  * Treatment level 2: Patients receive cetuximab, cisplatin, and radiotherapy as in treatment level 1. Patients also receive docetaxel IV over 1-2 hours once weekly in weeks 7-11.

Cohorts of 7-20 patients are treated at treatment level 1 or 2 sequentially, as long as no more than 2 of 7 patients experience dose-limiting toxicity (DLT), until the safe treatment level for future study is determined. The safe treatment level is defined as the level at which no more than 2 of 7 and no more than 6 of 20 patients experience DLT. At least 20 patients are treated at the safe treatment level.

* Surgery: Between 4-8 weeks after completion of neoadjuvant chemoimmunotherapy and radiotherapy, patients undergo surgery.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the thoracic esophagus

  * Carcinoma of the gastroesophageal junction (i.e., Siewert staging system type I disease) allowed
* Locally advanced disease

  * Obstructive tumors are considered locally advanced disease
  * Meets 1 of the following staging criteria:

    * T3, N0 disease
    * T1-3, N1 disease
    * T4, N0-1 disease
* Resectable disease

  * No T4 (unequivocal organ involvement) disease that cannot be resected with curative intent
* No airway infiltration in case of tumors of the upper third of the thoracic esophagus
* No cervical esophageal carcinoma
* No distant metastasis, including stage M1a (celiac node involvement) by fine-needle aspiration or biopsy

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Creatinine clearance > 60 mL/min
* Bilirubin normal
* Alkaline phosphatase ≤ 2.5 times upper limit of normal (ULN)
* AST ≤ 1.5 times ULN
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No other malignancy within the past 5 years except nonmelanomatous skin cancer or adequately treated in situ cervical cancer
* No severe or uncontrolled cardiovascular disease including, but not limited to, any of the following:

  * New York Heart Association class III or IV congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction within the past 3 months
  * Significant arrhythmias
* No psychiatric disorder that would preclude study compliance
* No active uncontrolled infection
* No serious underlying medical condition that, in the opinion of the investigator, would interfere with study participation (e.g., uncontrolled diabetes mellitus or active autoimmune disease)
* No peripheral neuropathy > grade 1
* No contraindications to corticosteroids
* No known hypersensitivity to any component of the study drugs

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior radiotherapy to the chest
* No participation in another clinical trial within the past 30 days
* No other concurrent experimental drugs or anticancer therapy
* No concurrent drugs contraindicated for use with the study drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Determine the safety of neoadjuvant radiotherapy in combination with cetuximab, docetaxel, and cisplatin | Until treatment ends
  Determine the safety of neoadjuvant radiotherapy in combination with cetuximab, docetaxel, and cisplatin

SECONDARY OUTCOMES:
Determine the feasibility and efficacy of the study's regimen | Until trial ends
  Determine the feasibility and efficacy of this regimen in these patients.
Determine the duration of response and patterns of failure | Until trial ends
  Determine the duration of response and patterns of failure in patients treated with this regimen

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ruhstaller, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (2):
- Switzerland (2):
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Klinik Stephanshorn, Sankt Gallen

REFERENCES:
- [Result] Ruhstaller T, Pless M, Dietrich D, Kranzbuehler H, von Moos R, Moosmann P, Montemurro M, Schneider PM, Rauch D, Gautschi O, Mingrone W, Widmer L, Inauen R, Brauchli P, Hess V. Cetuximab in combination with chemoradiotherapy before surgery in patients with resectable, locally advanced esophageal carcinoma: a prospective, multicenter phase IB/II Trial (SAKK 75/06). J Clin Oncol. 2011 Feb 20;29(6):626-31. doi: 10.1200/JCO.2010.31.9715. Epub 2011 Jan 4. PMID 21205757
- [Derived] Steffen T, Dietrich D, Schnider A, Kettelhack C, Huber O, Marti WR, Furrer M, Gloor B, Schiesser M, Thierstein S, Brauchli P, Ruhstaller T; Swiss Group for Clinical Cancer Research (SAKK). Recurrence Patterns and Long-term Results After Induction Chemotherapy, Chemoradiotherapy, and Curative Surgery in Patients With Locally Advanced Esophageal Cancer. Ann Surg. 2019 Jan;269(1):83-87. doi: 10.1097/SLA.0000000000002435. PMID 28742685